CLINICAL TRIAL: NCT06960239
Title: Evaluation of the Efficacy and Safety of an Irreversible Electroporation (IRE) System for The Treatment of Upper Airway Obstruction Due to Adenotonsillar Hypertrophy in Children
Brief Title: Safety and Efficacy of the Irreversible Electroporation (IRE) System for Adenotonsillar Hypertrophy in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ENTire Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN 0299
Record Dates: First submitted 2025-04-10; First posted 2025-05-07 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Tonsillar Hypertrophy; Upper Airway Obstruction
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Intervention Model Description: Irreversible Electroporation (IRE) System for the Treatment of Upper Airway Obstruction due to Adenotonsillar Hypertrophy in Children
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Enlarged tonsil(s) and/or adenoid mass will be reduced by ENTire IRE System. (Experimental): The bi-polar IRE System locally applies short, high-voltage (HV) pulses, increasing the permeability of tissue cells, creating non-thermal irreversible electroporation (NTIRE). The energy is transferred via bipolar forceps handpiece causing irreversible cell membrane perforation and apoptosis resulting in tissue reduction. The clinical effect is anticipated within 2 to 4 weeks post-treatment.
  Interventions: Device: IRE System

INTERVENTIONS:
Device: IRE System — Irreversible Electroporation (IRE) System for the Treatment of Upper Airway Obstruction due to Adenotonsillar Hypertrophy in Children
  Other Names: ENtire IRE System

SUMMARY:
This is a multi-center, prospective, open-label, traditional feasibility study with a before-after study design. The study is designed to evaluate the safety and efficacy of an Irreversible Electroporation (IRE) System for the treatment of upper airway obstruction due to adenotonsillar hypertrophy in Children.

DETAILED DESCRIPTION:
The purpose of the IRE System is to address the clinical need for reducing the volume of hypertrophic tonsil(s) and adenoid while minimizing side effects and complications. Procedure time will also be reduced. The IRE System is designed to be more comfortable for patients, as it employs a noninvasive procedure using a high voltage pulsed electric field to create irreversible nanopores in the cell membrane, leading to cell death and the reduction of the tonsils and adenoid volume. On basis of these finding and in view of the known safety profile and efficacy of current adeno-tonsillar reduction technologies, the purpose of the current study is to prospectively determine the efficacy and safety of the IRE System in adeno-tonsillar reduction.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 - 18 years.
* Tonsillar hypertrophy (more than 2 in Brodsky Grading System for Tonsils (BGST)).
* Symptomatic Upper Airway obstruction.

Exclusion Criteria:

* Age below 3 years, or above 18 years.
* Patients which underwent prior tonsillectomy or tonsillotomy.
* Body Mass Index (BMI) above the 95th percentile for patient's age and sex, as per the Centers for Disease Control and Prevention (CDC) growth charts.
* Patients with a pacemaker or similar electro stimulator implants.
* Patients for whom the anesthesia involves high risk.
* Epilepsy or other condition involving convulsions.
* Significant systemic illness (e.g., cancer, severe autoimmune disease, neurological disease).
* Bleeding diathesis.
* Known or suspected complications for any general or local anesthetic agents.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of days from treatment until no pain reported in Pain Scale. | 3 months post treatment
  The number of days from treatment until no pain is reported using the Wong-Baker FACES® Pain Scale is non-inferior to literature for other adenotonsillar surgeries. The Wong-Baker FACES® Pain Scale (Pain Scale) is a horizontal scale ranging from 0 "No hurt" to 10 "Hurts worst".
Evaluation of Sleep-Disordered Breathing | 3 months post treatment
  Obstructive Sleep Apnea (OSA) -18 questionnaire scoring change by 30% at 3 months compared to the Baseline. OSA -18 questionnaire includes 18 questions that rates the severity of different aspects of a child's life affected by OSA. Ratings are provided on a scale of 1 to 7, where a score of 1 refers to "None of the time" and a score of 7 "All of time". A final summed score could vary from 18 to 126, with higher scores indicating more severe symptoms and greater impairment.
Number of participants with treatment-related adverse events as assessed by a standardized 0-3 severity scale (0 = none, 1 = mild, 2 = moderate, 3 = severe). | 3 months post treatment
  Physician assessment of the incidence of post-treatment Adverse Events using a 0 to 3 grading scale (0=none, 1=mild, 2=moderate, 3=severe) following treatment and recording any additional side effects and comparing to literature for other adeno-tonsillar surgeries to check for non-inferiority.

SECONDARY OUTCOMES:
Sleep-Related Breathing Disorder Scale (PSQ-SRBD Scale) | 3 months post treatment
  Improvement in the PSQ-SRBD questionnaire score for Snoring, Sleeping and Behavior parameters, at 3 months compared to the Baseline. PSQ-SRBD scale contains 22 symptom items. Responses are "yes" = 1, "no" = 0, and "don't know"=missing. The mean response on non-missing items is the score, which can vary from 0 to 1.
  Higher scores suggest a higher risk for pediatric sleep-related breathing disorder.
Procedure Time | Intraoperative
  Procedure time reported is lower by 30% compared to literature for other adeno-tonsillar surgeries
Intraoperative blood loss | Intraoperative
  Intraoperative blood loss (mL)

CONTACTS AND LOCATIONS:
Locations (2):
- Spitalul Clinic de Urgență pentru copii "Maria S. Curie", Bucharest, Romania
- Republican Specialized Scientific-Practical Medical Center of Otorhinolaryngology and Head and Neck Diseases, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: No